CLINICAL TRIAL: NCT04363528
Title: Incidence of Deep Vein Thrombosis at Doppler Echo in Patients With SARS-Cov-2 Pneumopathy Hospitalized in ICU
Brief Title: Incidence of Deep Vein Thrombosis at Doppler Echo in Covid-19 Patients With SARS-Cov-2 Pneumopathy Hospitalized in ICU
Acronym: COVIDOP-DVT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Versailles Hospital (Other)
Responsible Party: Principal Investigator, Aurelien Maurizot, coordonator investigator, Versailles Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: P20/08_COVIDOP-DVT
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep Vein Thrombosis; doppler echo; SARS-CoV-2; ICU
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Doppler Echo (Other): patients will have a Doppler Echo when they enter ICU (within 48 hours) and a second Doppler Echo 7 days later
  Interventions: Other: Doppler Echo

INTERVENTIONS:
Other: Doppler Echo — 2 doppler echo will be done at patients hospitalized in ICU and with SARS-CoV-2 pneumopathy at 7 days apart

SUMMARY:
The main objective of the study is to determine the incidence of deep vein thromboses at Doppler echo in patients with SARS-Cov-2 pneumopathy upon their entry into ICU and after 7 days of hospitalization in ICU.

This is a monocentric interventional study (RIPH 2).

ELIGIBILITY:
Inclusion Criteria:

* Patient > or =18 years
* Hospitalization in intensive care
* PCR COVID 19+ or compatible clinical signs (fever, cough, myalgia, asthenia, loss of taste, anosmia) associated with compatible radiological signs

Exclusion Criteria:

* Pregnancy in progress
* Patient <18 years
* Patients deprived of freedoms or under guardianship
* Patient or family opponent of protocol participation
* patient on curative anticoagulant for more than 48H00
* impossible Venous Doppler Echo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2021-06-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Deep Vein Thrombosis at Doppler Echo in Patients With SARS-Cov-2 Pneumopathy Hospitalized in ICU | Day 0
  Deep vein thrombosis at Doppler echo
Incidence of Deep Vein Thrombosis at Doppler Echo in Patients With SARS-Cov-2 Pneumopathy Hospitalized in ICU | Day 7
  Deep vein thrombosis at Doppler echo

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de Versailles, Le Chesnay, France